CLINICAL TRIAL: NCT00006051
Title: Combination Chemotherapy Concurrent With Postoperative Radiotherapy Epidermoid Carcinoma of the Head and Neck at High Risk of Recurrence - Study of Feasibility
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068073; FRE-FNCLCC-GORTEC98-01/98007; EU-20015
Record Dates: First submitted 2000-07-05; First posted 2004-03-25 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one chemotherapy drug with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus radiation therapy in treating patients who have head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity of fluorouracil and cisplatin with concurrent radiotherapy in patients with stage I-IVB squamous cell cancer of the head and neck at high risk of recurrence following curative resection. II. Determine the efficacy of this regimen in these patients. III. Determine the survival of these patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients receive fluorouracil IV continuously on days 1-5 and 43-47 and cisplatin IV over 1 hour on days 2, 23, and 44. Concurrent radiotherapy is administered 5 days a week for 6.5 weeks. Patients are followed every 3 months for 2 years, then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 44-68 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage I-IVB squamous cell cancer of the oral cavity, oropharynx, hypopharynx, or larynx Positive lymph nodes allowed, either bilateral or contralateral Curatively resected within past 6 weeks No distant metastases

PATIENT CHARACTERISTICS: Age: Over 18 to 70 Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: WBC at least 2,000/mm3 Platelet count at least 150,000/mm3 Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) SGOT and SGPT less than 2 times ULN Alkaline phosphatase less than 2 times ULN Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance greater than 70 mL/min Cardiovascular: No contraindication to fluorouracil IV No coronary artery disease greater than grade 2 No unstable heart disease Other: No other malignancy except basal cell skin cancer or carcinoma in situ of the cervix Not pregnant Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics Other: No other concurrent adjuvant therapy No concurrent preventive treatment (e.g., retinoids) No other concurrent experimental treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-02 (Actual); Primary Completion 2002-08 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lionnel Geoffrois, MD, Study Chair — Centre Alexis Vautrin
Locations (6):
- France (6):
  - Centre Jean Perrin, Clermont-Ferrand
  - Hopital Jean Monnet, Épinal
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif